CLINICAL TRIAL: NCT04902144
Title: Breast and Ovarian Catchment Pilot Grant: Clinical Outcomes for Offering Genetic Testing in a Tiered Approach
Brief Title: Clinical Outcomes for Offering Genetic Testing in a Tiered Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Marianne Dubard-Gault, Assistant Professor, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: RG1121550; NCI-2021-04181 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00010137 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2021-05-17; First posted 2021-05-26 (Actual); Results first posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Breast Carcinoma; Colon Carcinoma; Malignant Solid Neoplasm; Ovarian Carcinoma; Pancreatic Carcinoma; Prostate Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening (medical records, coaching) (Experimental): PHASE I: Patients' medical data are collected.
  PHASE II: Patients complete questionnaires and their medical data is collected. SCCA subject matter experts and OMC providers review patients' medical data at bi-monthly virtual conferences. OMC providers receive coaching from SCCA subject matter experts for guidance on providing genetic counseling and testing to their patients.
  Interventions: Other: Electronic Health Record Review; Other: Questionnaire Administration; Behavioral: Behavioral Intervention

INTERVENTIONS:
Other: Electronic Health Record Review — Medical data collected
Other: Questionnaire Administration — Complete questionnaires
Behavioral: Behavioral Intervention — Receive coaching
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments

SUMMARY:
This clinical quality improvement study reviews and develops a clinical operations workflow to identify cancer patients who meet criteria for genetic counseling and testing. This study may improve utilization of genetic counseling and testing amongst community-based oncology providers caring for cancer patients in a rural and underserved area.

DETAILED DESCRIPTION:
OUTLINE: Medical oncologists at Olympic Medical Center (OMC) participated in this study and received a peer coaching intervention during phase II to help identify patients who meet criteria for genetic counseling and testing

PHASE I: Patients' medical data are collected; no intervention.

PHASE II: Olympic Medical Center (OMC) patients complete family history questionnaires and their medical data are collected. Seattle Cancer Care Alliance (SCCA) subject matter experts and OMC providers review patients' medical data at bi-weekly virtual conferences. OMC providers will be consenting to release their patients' medical records to SCCA so that SCCA subject matter experts (cancer geneticist and/or genetic counselor) can identify patients with an underlying hereditary cancer syndrome to be offered genetic counseling and testing.

OMC providers receive coaching from SCCA subject matter experts for guidance on providing genetic counseling and testing to their patients.

ELIGIBILITY:
Inclusion Criteria:

* Medical oncology providers at OMC who see patients with an active diagnosis of breast, ovarian, prostate, colon, or pancreatic cancer

Exclusion Criteria:

* OMC providers who do not see patients with an active diagnosis of cancer
* OMC providers who see patients who are minors
* OMC providers who see patients with precancerous lesions such as ductal carcinoma in situ (the presence of abnormal cells inside a milk duct in the breast) or colon polyps (a small clump of cells that form on the lining of the colon or rectum)

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Dubard-Gault, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Olympic Medical Cancer Center, Sequim, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Medical Data Collection, Peer Coaching: PHASE I: Patients' medical data are collected,
  PHASE II: Olympic Medical Center (OMC) patients complete family history questionnaires and their medical data are collected. Seattle Cancer Care Alliance (SCCA) subject matter experts and OMC providers review patients' medical data at bi-weekly virtual conferences. OMC providers will be consenting to release their patients' medical records to SCCA so that SCCA subject matter experts (cancer geneticist and/or genetic counselor) can identify patients with an underlying hereditary cancer syndrome to be offered genetic counseling and testing.
  OMC providers receive coaching from SCCA subject matter experts for guidance on providing genetic counseling and testing to their patients.
  Electronic Health Record Review: Medical data collected
  Questionnaire Administration: Complete questionnaires
Period: Overall Study
Arm/Group | Medical Data Collection, Peer Coaching
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Medical Data Collection, Peer Coaching
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 55 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Identify Cancer Patients Who Meet Criteria for Genetic Counseling and Testing
Description: The number of cancer patients who meet criteria for genetic counseling and testing as identified by the study team and OMC oncology providers
Time Frame: 6 months
Measure: Number; unit: patients
Groups:
- Medical Data Collection Without Peer Coaching: PHASE I: Medical oncologists enrolled, Patients' medical data are collected but were not enrolled.
- Medical Data Collection With Peer Coaching: PHASE II: Olympic Medical Center (OMC) patients complete family history questionnaires and their medical data are collected, they were not enrolled. medical oncologists seeing them were enrolled as participants. Seattle Cancer Care Alliance (SCCA) subject matter experts and OMC providers review patients' medical data at bi-weekly virtual conferences. OMC providers will be consenting to release their patients' medical records to SCCA so that SCCA subject matter experts (cancer geneticist and/or genetic counselor) can identify patients with an underlying hereditary cancer syndrome to be offered genetic counseling and testing.
  OMC providers receive coaching from SCCA subject matter experts for guidance on providing genetic counseling and testing to their patients.
  Electronic Health Record Review: Medical data collected Questionnaire Administration: Complete questionnaires
Arm/Group | Medical Data Collection Without Peer Coaching | Medical Data Collection With Peer Coaching
Number analyzed (Participants) | 6 | 6
patients | 100 | 48

2. Primary Outcome: Uptake of Genetic Testing
Description: Number of genetic testing ordered and processed for patients with cancer who meet criteria for testing. Out of 415 patients seen in phase I, 100 met criteria but only 29 received testing. Out of 219 patients seen in phase II, 48 met criteria but only 25 received testing.
Time Frame: Up to study completion (Assessed up to1 year and 4 months)
Population: The number of genetic testing kits ordered and processed for patients with cancer who meet criteria for testing in phase I and phase II
Measure: Number; unit: tests
Arm/Group | Medical Data Collection Without Peer Coaching | Medical Data Collection With Peer Coaching
Number analyzed (Participants) | 415 | 219
tests | 29 | 25

3. Primary Outcome: Clinical and Patient Reported Outcomes Following Genetic Test Results
Description: Pertinent clinical information regarding genetic test result and related outcomes (referrals, treatment recommendations); pulled directly from electronic health record, genetic test reports, and patient questionnaires
Time Frame: Up to study completion (Assessed up to 1 year and 4 months)
Population: 5 patients were referred to our center for post test counseling and treatment recommendations in the setting of positive results. Many other patients could have chosen to go to a cancer genetic clinic closer to their home.
Measure: Count of Participants; unit: Participants
Arm/Group | Medical Data Collection Without Peer Coaching | Medical Data Collection With Peer Coaching
Number analyzed (Participants) | 415 | 219
Participants | 2 | 3

ADVERSE EVENTS:
Time Frame: Adverse events were not collected for this study
Description: This study did peer coaching of medical oncologists as study participants. No patients were considered study participants. Adverse events were not collected for this study.
Groups:
- Screening (Medical Records, Coaching): PHASE I: Patients' medical data are collected.
  PHASE II: Patients complete questionnaires and their medical data is collected. SCCA subject matter experts and OMC providers review patients' medical data at bi-monthly virtual conferences. OMC providers receive coaching from SCCA subject matter experts for guidance on providing genetic counseling and testing to their patients.
  Electronic Health Record Review: Medical data collected
  Questionnaire Administration: Complete questionnaires
  Behavioral Intervention: Receive coaching
Arm/Group | Screening (Medical Records, Coaching)
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
This study was not a clinical trial, it was a quality improvement project of practices of rural medical oncologists to increase their ordering of GT when indicated for their patients with active cancer. Six rural oncologists participated in both phases, the observation phase and the peer coaching phase, and and for the full length of QI study. Number of patients seen and number of tests ordered was collected to measure effectiveness of peer coaching. No data on adverse events were collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/44/NCT04902144/Prot_001.pdf
  • Informed Consent Form (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/44/NCT04902144/ICF_002.pdf